CLINICAL TRIAL: NCT05432141
Title: Safety Observation of Sabin Inactivated Poliovirus Vaccine (Vero Cell) in Primary Immunization, Booster Immunization and Simultaneous Vaccination With Other Vaccines in Infants
Brief Title: A Safety Study of Sabin Inactivated Poliovirus Vaccine in Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-sIPV-MA4001-JX
Record Dates: First submitted 2022-06-20; First posted 2022-06-27 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-06

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis | interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines; Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary immunization group (Experimental): A total of 2000 infants aged 2-3 months will randomly assigned to two groups according to 1:1 using scratch cards: 1000 infants in the sIPV vaccine group and 1000 infants in the sIPV vaccine group plus DTaP vaccine group
  Interventions: Biological: sIPV vaccine /DTaP vaccine
- Booster immunization group of sIPV vaccine (Experimental): A total of 1200 children aged 18 months will randomly assigned to four groups according to 2:2:1:1 using scratch cards: 400 in the sIPV booster group, 400 in the sIPV booster group plus inactivated hepatitis A vaccine simultaneously, 200 in the sIPV booster group plus MMR simultaneously, and 200 in the sIPV booster group plus attenuated hepatitis A vaccine.
  Interventions: Biological: sIPV vaccine /Hepatitis A inactivated vaccine /MMR vaccine

INTERVENTIONS:
Biological: sIPV vaccine /DTaP vaccine — All subjects received 3 doses of sIPV vaccines and 3 doses of DTaP vaccines. Subjects recommended intramuscular injection. The best site for intramuscular injection is the anterolateral middle thigh for infants and the deltoid muscle for children.
  Arms: Primary immunization group
Biological: sIPV vaccine /Hepatitis A inactivated vaccine /MMR vaccine — All subjects will receive 1 dose of sIPV and 2 doses of hepatitis A inactivated vaccine/or 1 dose of attenuated hepatitis A vaccine and 1 dose of MMR vaccine.Subjects recommended intramuscular injection. The best site for intramuscular injection is the anterolateral middle thigh for infants and the deltoid muscle for children.
  Arms: Booster immunization group of sIPV vaccine

SUMMARY:
The purpose of this study is to evaluate the safety of Sabin Inactivated Poliovirus Vaccine (Vero cell)(sIPV)in the primary immunization of infants at the age of 2 months and booster immunization of children at the age of 18 months, and the simultaneous immunization with other vaccines of children at the age of 2 months and older, so as to provide reference for the improvement of immunization strategy.

DETAILED DESCRIPTION:
This study is an open and observational phase Ⅳ clinical trial of Sabin Inactivated Poliovirus Vaccine.The purpose of this study is to evaluate the safety of Sabin Inactivated Poliovirus Vaccine (Vero cell)(sIPV)in the primary immunization of infants at the age of 2 months and booster immunization of children at the age of 18 months, and the simultaneous immunization with other vaccines of children at the age of 2 months and older, so as to provide reference for the improvement of immunization strategy.A total of 3200 subjects including 2000 subjects aged 2~3 months in primary immunization group,1200 subjects aged 18 months in primary immunization group will be enrolled and will receive sIPV vaccine or sIPV vaccine and other vaccines simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 2-3 months should be involved in primary immunization and they have not received Sabin strain inactivated polio vaccine (Vero Cell) in the past;
* Children aged 18 months should be immunized with the first three doses of Sabin strain inactivated polio vaccine (Vero Cell) and they have not received any inactivated or attenuated live vaccines in the past 14 days;
* The guardian agrees to sign the informed consent and voluntarily use the mobile APP to participate in the follow-up visits.

Exclusion Criteria:

* Allergic to the active ingredient in the vaccine, any inactive ingredient, or substance used in the manufacturing process;
* Allergic to this product or similar vaccines in the past;
* Patients with severe chronic diseases or allergies;
* Patients with fever or acute illness.

The Exclusion Criteria for the Second and Third Doses:

* Any serious adverse events that are causally related to vaccination;
* Severe anaphylaxis or hypersensitivity after vaccination (including hives and rashes within 30 minutes of vaccination);
* Any confirmed or suspected autoimmune or immunodeficiency disease, including human immunodeficiency virus (HIV) infection;
* Acute or newly emerging chronic diseases occur at the time of vaccination;
* Other reactions (including severe pain, severe swelling, severe limitation of movement, persistent high fever, severe headache, or other systemic or local reactions), as determined by the investigator;
* Having an acute illness at the time of vaccination (acute illness is defined as moderate or severe illness with or without fever);
* Axillary temperature >37℃ during vaccination.

Ages: 2 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3200 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reactions within 0~7 days after primary immunization of sIPV vaccine | Within 0~7 days after primary immunization
  Incidence of adverse reactions within 0~7 days after primary immunization of sIPV vaccine

SECONDARY OUTCOMES:
Incidence of adverse reactions within 0~30 days after primary immunization of sIPV vaccine | Within 0~30 days after primary immunization
  Incidence of adverse reactions within 0~30 days after primary immunization of sIPV vaccine.
Incidence of adverse reactions within 0~7 days after booster immunization of sIPV vaccine | Within 0~7 days after booster immunization
  Incidence of adverse reactions within 0~7 days after booster immunization of sIPV vaccine .
Incidence of adverse reactions within 0~30 days after booster immunization of sIPV vaccine | Within 0~30 days after booster immunization
  Incidence of adverse reactions within 0~30 days after booster immunization of sIPV vaccine.
Incidence of adverse reactions within 0-7 days after primary immunization of sIPV vaccine combined with DTaP vaccine | Within 0-7 days after primary immunization combined with DTaP vaccine
  Incidence of adverse reactions within 0-7 days after primary immunization of sIPV vaccine combined with DTaP vaccine.
Incidence of adverse reactions within 0-30 days after primary immunization of sIPV vaccine | Within 0-30 days after primary immunization combined with DTaP vaccine
  Incidence of adverse reactions within 0-30 days after primary immunization of sIPV vaccine combined with DTaP vaccine.
Incidence of adverse reactions after booster immunization of sIPV vaccine combined with inactivated hepatitis A vaccine | Within 0~7 days after booster immunization combined with inactivated hepatitis A vaccine
  Incidence of adverse reactions within 0~7 days after booster immunization of sIPV vaccine combined with inactivated hepatitis A vaccine.
Incidence of adverse reactions within 0 ~14 days after booster immunization of sIPV vaccine | Within 0 ~14 days after booster immunization
  Incidence of adverse reactions within 0 ~14 days after booster immunization of sIPV vaccine combined with MMR vaccine or attenuated hepatitis A vaccine.
Incidence of adverse events within 0 ~ 30 days after booster immunization of sIPV vaccine | Within 0 ~ 30 days after booster immunization of sIPV vaccine combined with MMR vaccine ,inactivated hepatitis A vaccine or attenuated hepatitis A vaccine.
  Incidence of adverse events within 0 ~ 30 days after booster immunization of sIPV vaccine combined with MMR vaccine ,inactivated hepatitis A vaccine or attenuated hepatitis A vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Shicheng Guo, Master, Principal Investigator — Jiangxi Provincial Center for Disease Prevention and Control
Locations (2):
- China (2):
  - Gaoan Center for Disease Control and Prevention, Gao’an, Jiangxi
  - Shangli County Center for Disease Control and Prevention, Pingxiang, Jiangxi

REFERENCES:
- [Derived] Guo S, Li Z, Zheng M, Wu F, Sun J, Tuo L, Li S, Li X, Wei L, Xia Z, Xie P, Chen X, Zhao Y, Gao Y, Yu D. Safety and 6-month immune persistence of inactivated poliovirus vaccine (Sabin strains) simultaneously administrated with other vaccines for primary and booster immunization in Jiangxi Province, China. Vaccine. 2024 Aug 30;42(21):126183. doi: 10.1016/j.vaccine.2024.126183. Epub 2024 Jul 31. PMID 39088987